CLINICAL TRIAL: NCT02799680
Title: Treatment of Relapsed and/or Refractory CD33-positive Acute Myeloid Leukemia by Infusions of Allogeneic CART-33
Brief Title: Allogeneic CART-33 for Relapsed/Refractory CD33+ AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-AML-2015
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Relapsed and/or Refractory CD33+ AML
Keywords: CART; AML

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogeneic CART-33 (Experimental): infusions of allogeneic CD33-directed chimeric antigen receptor-modified T cells (CART-33)
  Interventions: Biological: allogeneic CART-33

INTERVENTIONS:
Biological: allogeneic CART-33 — allogeneic CD33-directed chimeric antigen receptor-modified T cells (CART-33)

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of allogeneic cluster of differentiation 33 (CD33)-directed chimeric antigen receptor modified T cells (CART-33) infusions in patients with relapsed / refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The relapsed and/or refractory AML patients will receive infusions of allogeneic CART-33 within 1 week after chemotherapy. The re-induction chemotherapy regimen was primarily idarubicin and cytarabine, and no graft-versus-host disease (GVHD) prevention was conducted pre- and post- therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Patient with relapsed and/or refractory CD33 positive acute myeloid leukemia (AML)
* Estimated life expectancy ≥ 12 weeks (according to investigator's judgment)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Previous treatment with investigational gene or cell therapy medicine products
* CD33 negative leukemia
* Any uncontrolled active medical disorder that would preclude participation as outlined
* Pregnant or lactating women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 1 year
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria

SECONDARY OUTCOMES:
Overall response rate of allogeneic CART-33 | up to 24 weeks
  A response is defined as: (1) a morphologic complete remission (CR) or (2) a complete remission with incomplete recovery of counts (CRi) (based on NCCN guidelines (National Comprehensive Cancer Network (NCCN), 2015) or (3) a negative minimal residual disease assessed by flow cytometry or qPCR
Disease-free survival | up to 24 weeks
Overall survival | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Ai, MD, Study Chair — Affiliated Hospital of Academy of Military Medical Sciences
Locations (2):
- China (2):
  - Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided